CLINICAL TRIAL: NCT07237022
Title: The Role of Transient Receptor Potential Channels in Diabetic Peripheral Neuropathy
Brief Title: The Role of TRP Channels in DPN
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: CCP24-3303-DPN
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-06

CONDITIONS: Physiological Responses
MeSH Terms: interventions — cinnamaldehyde; allyl isothiocyanate; Capsaicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cinnamaldehyde — A 10% and 30% cinnamaldehyde solution is topically applied on foot skin.
Other: Allyl isothiocyanate (AITC) — A 15% and up to 30% AITC solution is topically applied on foot skin.
Other: Capsaicin — A 1.5% and 5% capsaicin solution is topically applied on foot skin.

SUMMARY:
The study aims to characterize the vascular response upon topical application of cinnamaldehyde, allyl isothiocyanate and capsaicin on feet skin in healthy volunteers. The vascular response will be characterized in terms of response over time, dose-response, inter-foot and inter-period reproducibility.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a white male or female ≥18 and ≤45 years of age
2. Subject is a non-smoker for at least 6 months prior to the start of the study
3. Subject has a body mass index (BMI) between 18-30 kg/m²
4. Subject is judged to be in good general health on the basis of medical history, physical examination and vital signs
5. Subject understands the procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

1. Subject has a history of any illness or disorder which, in the investigator's opinion, might confound the results of the study
2. Subject has a history of significant severe (drug) allergies
3. Subject is a female who is pregnant, breast-feeding or intends to become pregnant, or is of child-bearing potential and is not using an adequate contraceptive method
4. Subject uses any prescription or non-prescription drugs on a regular basis which, in the investigator's opinion, might confound the results of the study
5. Subject currently uses lotions, oils, depilatory preparations, makeup, or other topical treatments on the feet on a regular basis which cannot be discontinued for the duration of the study
6. Subject has eczema, scleroderma, psoriasis, dermatitis or keloids, tumors, ulcers, burns, skin flaps or grafts on the volar surface of the forearm or the dorsum of the feet, or any other skin abnormality that, in the opinion of the investigator, may interfere with the study assessments
7. Subject has excessive hair growth on the volar surface of the forearms or the dorsum of the feet
8. Subject has any of the following vital sign measurements at screening after at least 10 minutes of supine rest: Heart Rate <40 or >100 beats/min, Diastolic Blood Pressure <50 or >90 mmHg, Systolic Blood Pressure <90 or >140 mmHg
9. Subject is unable to refrain from drinking caffeinated beverages (e.g. coffee, tea, cola, …) 24 hours prior to each study visit. Subject is unable to limit their intake of caffeinated beverages to ≤4 cups a day throughout the study
10. Subject is unable to refrain from drinking alcohol 24 hours prior to each study visit, is currently a regular user of illegal drugs, or has a history of substance abuse (including alcohol)
11. Subject is currently participating or has been involved in testing an investigational drug in another clinical study within the last 4 weeks
12. Subject is in a situation or has a condition which, in the opinion of the investigator, may interfere with safe and optimal participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy male and female volunteers aged 18 to 45 years (inclusive)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Dermal Blood Flow response (PU) | Up until 60 minutes after cinnamaldehyde and AITC application; and up until 90 minutes after capsaicin application.
  The DBF response prior to and at each point in time after topical application of cinnamaldehyde, AITC and capsaicin on the foot, assessed with LSCI, within the area of application, expressed in arbitrary perfusion units (PU).
Flare area (mm²) | Up until 60 minutes after cinnamaldehyde and AITC application; and up until 90 minutes after capsaicin application.
  The flare area of the DBF response prior to and at each point in time after topical application of cinnamaldehyde, AITC and capsaicin on the feet, assessed with LSCI.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) pain score | Up until 60 minutes after cinnamaldehyde and AITC application; and up until 90 minutes after capsaicin application.
  The Numeric Rating Scale (NRS)-11 pain score at each point in time after topical application of cinnamaldehyde, AITC and capsaicin on the feet.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Pharmacology, Leuven, Belgium